CLINICAL TRIAL: NCT03265886
Title: The Influence of Bupivacaine Temperature on Supraclavicular Plexus Block Characteristics
Brief Title: The Influence of Warm Bupivacaine on Supraclavicular Plexus Block Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MFM-IRB, MS/17.05.143
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Surgery to the Distal One Third of the Upper Limb

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double-blind design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm bupivacaine at (37°c) (Experimental): Warmed bupivacaine at body temperature will be administered
  Interventions: Drug: Warm bupivacaine at (37°c)
- Bupivacaine at operating room temperature (23°c) (Active Comparator): Bupivacaine at temperature of 23°C will be administered
  Interventions: Drug: Bupivacaine at operating room temperature (23°c)

INTERVENTIONS:
Drug: Warm bupivacaine at (37°c) — Bupivacaine 0.5%, 30 mL, warmed to 37◦C for 20 minutes. The empty syringes and needles, in their packaging, will be held at the same temperature before initiating the block.
  Arms: Warm bupivacaine at (37°c)
Drug: Bupivacaine at operating room temperature (23°c) — Bupivacaine 0.5%, 30 ml held in crash shelf of the operating room temperature at 23◦C. The empty syringes and needles will be held in the same temperature before use.
  Arms: Bupivacaine at operating room temperature (23°c)

SUMMARY:
Despite PH adjustment of local anesthetic solution improves the quality of the block in all respects with special advantage of early onset of sensory and motor block, adequate level of analgesia, and prolongation of duration of block, the effect of warmed bupivacaine should have the same effect which have not been evaluated on supraclavicular plexus block for upper limb surgery.

The warmed bupivacaine used in supraclavicular plexus block may reduce sensory and motor block onset and prolong the duration of analgesia when compared to bupivacaine at operating room temperature.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of warm bupivacaine 0.5% at 37◦C versus bupivacaine 0.5% at operating room temperature at 23◦C on ultrasound-guided supraclavicular plexus block characteristics as regard sensory block onset time, motor block onset time, duration of sensory and motor block , effective duration of analgesia, total analgesics requirement, complications and side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I or II

Exclusion Criteria:

* Patient refusal.
* Pregnancy
* Neuromuscular diseases (as myopathies, myasthenia gravies…)
* Hematological diseases
* Bleeding disorders
* Coagulation abnormality.
* Psychiatric diseases.
* Local skin infection
* Sepsis at site of the block.
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2.
* Bilateral upper limb injury to be performed at the same procedure.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Time to onset of sensory block | for 30 min following injection
  defined as the time interval between the end of local anesthetic injection and the loss of sensation to pinprick (sensory score = 1)

SECONDARY OUTCOMES:
Time to onset of motor block | For 3 hours after the injection of local anesthetic
  defined as time interval between the end of local anesthetic injection and (motor score = 1) in the distributions of all 4 peripheral nerves.
Heart rate | For 3 hours after the injection of local anesthetic
Blood pressure | For 3 hours after the injection of local anesthetic
oxygen saturation in the peripheral blood | For 3 hours after the injection of local anesthetic
Duration of sensory block | For 24 hours after the injection of local anesthetic
  defined as the interval between end of injection and complete end of sensory block (score=2)
Duration of motor block | For 24 hours after the injection of local anesthetic
  defined as the interval between end of injection and complete recovery of normal motor function (score=0), respectively.
The severity of postoperative pain | For 24 hours after the injection of local anesthetic
  will be measured and recorded by using a 100-cm visual analog scale (VAS) for pain, where 0 is equal to no pain and 100 indicates the worst possible pain.
Time for first analgesic request | For 24 hours after the injection of local anesthetic
  Time to the first receiving of rescue analgesic from the time of blockade
Total analgesics received | for 24 hrs after the injection of local anesthetic
  Cumulative use of rescue analgesics after performing the blockade
Satisfaction Score | for 48 hrs after the injection of local anesthetic
  Using score including 5-Excellent, 4-Very Good, 3-Good, 2-Fair, and 1-Poor

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Y Makharita, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Faculty of Medicine, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
do not mind sharing raw data but after its publication not before.
Supporting Information: Study Protocol, SAP, ICF